CLINICAL TRIAL: NCT00929695
Title: A Phase III Study to Determine Efficacy and Safety of Low-Dose Glucocorticoids for Initial Treatment of Acute Graft-versus-Host Disease
Brief Title: Low-Dose Prednisone or Methylprednisolone in Treating Patients With Newly Diagnosed Acute Graft-versus-Host Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marco Mielcarek, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2327.00; NCI-2010-00323 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA018029 (NIH)
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Graft Versus Host Disease; Recurrent Adult Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Graft vs Host Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Prednisone; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate

ARMS (2):
- Arm I (Low-dose) (Experimental): Patients receive low-dose prednisone or methylprednisolone once or twice daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: prednisone; Drug: methylprednisolone; Other: questionnaire administration
- Arm II (Standard-dose) (Active Comparator): Patients receive standard-dose prednisone or methylprednisolone once or twice daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: prednisone; Drug: methylprednisolone; Other: questionnaire administration

INTERVENTIONS:
Drug: prednisone — immunosuppressive drug
  Other Names: DeCortin; Deltra
Drug: methylprednisolone — immunosuppressive drug
  Other Names: Depo-Medrol; Medrol; MePRDL; Solu-Medrol; Wyacort
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized phase III trial is studying low-dose prednisone or methylprednisolone to see how well they work compared with standard-dose prednisone or methylprednisolone in treating patients with newly diagnosed acute graft-versus-host disease (GVHD). Glucocorticoids, such as prednisone or methylprednisolone at a starting dose of 2 mg/kg/day are standard treatment for acute graft-versus-host disease caused by a donor stem cell transplant. It is not yet known whether low-dose glucocorticoids are more effective than standard-dose glucocorticoids in treating acute graft-versus-host-disease

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine whether a lower starting dose of prednisone for treatment of newly diagnosed acute GVHD results in decreased prednisone exposure without compromising overall survival.

II. To estimate the magnitude of clinical benefit associated with the reduction in prednisone exposure.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (Low-dose; prednisone-equivalent dose at initiation of treatment of 0.5 mg/kg/day or 1.0 mg/kg/day; stratified according to initial symptom severity): Patients receive low-dose prednisone or methylprednisolone once or twice daily in the absence of disease progression or unacceptable toxicity.

ARM II (Standard-dose; prednisone-equivalent dose at initiation of treatment of 1.0 mg/kg/day or 2.0 mg/kg/day; stratified according to initial symptom severity): Patients receive standard-dose prednisone or methylprednisolone once or twice daily in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 year and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed acute GVHD (>= grade IIa) for whom, in the judgment of the attending physician, initial treatment with systemic glucocorticoids is indicated
* Patient or guardian able and willing to provide informed consent

Exclusion Criteria:

* Hallmarks of chronic GVHD
* GVHD after donor lymphocyte infusion (DLI)
* Patient unwilling to remain in Seattle under the care of the Fred Hutchinson Cancer Research Center (FHCRC)/Seattle Cancer Care Alliance (SCCA) through day 42 after the start of treatment for GVHD
* Uncontrolled infection or other underlying comorbidity (i.e. severe psychiatric illness) that precludes the use of "standard-dose" prednisone
* Recent diagnosis of recurrent or progressive malignancy that precludes the use of "standard-dose" prednisone
* Any prior systemic therapy for acute GVHD (Patients may receive up to 2 doses of low-dose prednisone prior to randomization; low-dose prednisone is defined as 0.5 mg/kg/dose for patients who present with grade IIa GVHD and 1 mg/kg/dose for those who present with grade IIb-IV GVHD)
* Enrollment on Blood and Marrow Transplant Clinical Trials Network (BMT-CTN) trial 0802

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2009-06; Primary Completion 2013-07 (Actual); Study Completion 2015-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Mielcarek, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (Low-dose): Patients received prednisone-equivalent low doses of prednisone depending on presenting grade of acute GVHD (0.5 mg/kg/day for mild GVHD or 1.0 mg/kg/day for moderate/severe GVHD). Patients could receive prednisone or methylprednisolone.
- Group B (Standard-dose): Patients received prednisone-equivalent standard doses of prednisone depending on presenting grade of acute GVHD (1.0 mg/kg/day for mild GVHD or 2.0 mg/kg/day for moderate/severe GVHD). Patients could receive prednisone or methylprednisolone.
Period: Overall Study
Arm/Group | Group A (Low-dose) | Group B (Standard-dose)
Started | 81 | 83
Completed | 73 | 77
Not Completed | 8 | 6
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — discharge home | 4 | 3
Not completed — incorrect stratification | 2 | 0

BASELINE CHARACTERISTICS:
Population: From a total enrollment of 164 patients, 150 were analyzed for the primary endpoint. Excluded from the analysis were 14 patients: 12 withdrew, died or were discharged from the Center early and did not have 42 days of cumulative prednisone dosing and 2 were stratified incorrectly.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Low-dose) | Group B (Standard-dose) | Total
Number analyzed (Participants) | 73 | 77 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 14 | 22
  Between 18 and 65 years | 59 | 56 | 115
  >=65 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 26 | 57
  Male | 42 | 51 | 93

OUTCOME MEASURES:

1. Primary Outcome: Mean Cumulative Prednisone Dose (mg/kg) Over 42 Days From the Start of Treatment
Description: The total cumulative dose of prednisone (milligrams/kilogram) was calculated starting from the start of therapy through study day 42.
Time Frame: At day 42 after initiation of treatment
Population: From a total enrollment of 164 patients, the cumulative dose of prednisone at day 42 of treatment was available in 152 patients. The primary outcome was not measured in 12 patients due to withdrawal from study (2), discharge from Center before day 42 of treatment (10). Analysis was not completed in two patients due to an error in stratification.
Measure: Mean (Standard Deviation); unit: milligrams per kilogram
Groups:
- Grade IIa GVHD; 0.5 mg/kg/d Prednisone: Patients with mild acute GVHD were treated with a prednisone-equilavent dose of 0.5 mg/kg/day (low dose). Patients could be treated with prednisone or methylprednisolone.
- Grade IIa GVHD; 1.0 mg/kg/d Prednisone: Patients with mild acute GVHD were treated with a prednisone-equilavent dose of 1.0 mg/kg/day (standard dose). Patients could be treated with prednisone or methylprednisolone.
- Grade IIb-IV GVHD; 1.0 mg/kg/d Prednisone: Patients with moderate/severe acute GVHD were treated with a prednisone-equilavent dose of 1.0 mg/kg/day (low dose). Patients could be treated with prednisone or methylprednisolone.
- Grade IIb-IV GVHD; 2.0 mg/kg/d Prednisone: Patients with moderate/severe acute GVHD were treated with a prednisone-equilavent dose of 2.0 mg/kg/day (standard dose). Patients could be treated with prednisone or methylprednisolone.
Arm/Group | Grade IIa GVHD; 0.5 mg/kg/d Prednisone | Grade IIa GVHD; 1.0 mg/kg/d Prednisone | Grade IIb-IV GVHD; 1.0 mg/kg/d Prednisone | Grade IIb-IV GVHD; 2.0 mg/kg/d Prednisone
Number analyzed (Participants) | 44 | 47 | 29 | 30
milligrams per kilogram | 22.2 (13.7) | 27.1 (12.7) | 38.4 (14.1) | 41.3 (12.1)
Statistical Analysis 1: Comparison: Grade IIa GVHD; 0.5 mg/kg/d Prednisone vs Grade IIa GVHD; 1.0 mg/kg/d Prednisone; Test type: Superiority or Other; p = 0.08, t-test, 2 sided
Statistical Analysis 2: Comparison: Grade IIb-IV GVHD; 1.0 mg/kg/d Prednisone vs Grade IIb-IV GVHD; 2.0 mg/kg/d Prednisone; Test type: Superiority or Other; p = 0.4, t-test, 2 sided

2. Secondary Outcome: Prednisone-associated Toxicity as Assessed by Hyperglycemia
Description: Impact on blood glucose (BG) control will be assessed by comparing average BG and BG-variability between patients given standard-dose and low-dose prednisone.
Time Frame: Baseline and then through 42 days after starting treatment
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Group A (Low-dose) | Group B (Standard-dose)
Number analyzed (Participants) | 79 | 83
mg/dL | 140 (7.4) | 142 (12.9)

3. Secondary Outcome: Prednisone-associated Toxicity as Assessed by Invasive Infections (Bacterial, Fungal and Viral)
Description: The total number of invasive infections (bacterial, fungal and viral) occurring in patients in each group were collected.
Time Frame: Baseline and through 100 days of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Group A (Low-dose) | Group B (Standard-dose)
Number analyzed (Participants) | 79 | 83
percentage of participants | 52 | 53

4. Secondary Outcome: Prednisone-associated Toxicity as Assessed by Myopathy
Description: Assessed by mean change from baseline to day 42 using Manual Muscle Testing measure. The degree of resistance against pressure applied by tester was measured on a 5-point scale. A score of 5 indicates the patient can hold the position against maximum to strong resistance. A score of 0 indicates the patient has no resistance against pressure. Testing included upper and lower extremities: shoulder (deltoid at 90 degrees), and hip and knee in a sitting position.
Time Frame: Baseline and then weekly until 42 days after starting treatment
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Group A (Low-dose) | Group B (Standard-dose)
Number analyzed (Participants) | 79 | 83
units on a scale | -0.18 [-1.5 to 1.5] | -0.18 [-1.5 to 1.5]

5. Secondary Outcome: Prednisone-associated Toxicity as Assessed by Hypertension
Description: The number of different anti-hypertensive medications administered to control hypertension were collected. The mean change in the number of medications from baseline to day 42 was measured.
Time Frame: Baseline and then through 42 days after starting treatment
Measure: Mean (Full Range); unit: medications
Arm/Group | Group A (Low-dose) | Group B (Standard-dose)
Number analyzed (Participants) | 79 | 83
medications | -0.29 [-0.50 to 0.50] | -0.24 [-0.50 to 0.50]

6. Secondary Outcome: Prednisone-associated Toxicity as Assessed by Quality of Life
Description: Patients completed the MD Anderson Symptom Inventory (MDASI), which is a quality of life questionnaire validated for oncology/transplant patients. On a 1-10 point scale, patients scored the degree of severity of symptoms or the degree of interference in feelings or function due to symptoms at baseline or in the previous week. A score of 1 indicates symptom is not present or does not interfere with feelings or function. A score of 10 indicates the symptom is as bad as you can imagine or interferes completely with feelings or function. The mean change in score from baseline to day 42 was measured.
Time Frame: Baseline and then every other week until 42 days after starting treatment
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Group A (Low-dose) | Group B (Standard-dose)
Number analyzed (Participants) | 79 | 83
units on a scale | -2.3 [-5 to 5] | -1.9 [-5 to 5]

7. Secondary Outcome: Non-relapse Mortality
Description: Non-relapse mortality (NRM) is defined as death due to any cause in the absence of documented relapse/progression.
Time Frame: At 12 months after the start of prednisone therapy
Measure: Number; unit: percentage of participants
Arm/Group | Group A (Low-dose) | Group B (Standard-dose)
Number analyzed (Participants) | 79 | 83
percentage of participants | 15 | 16

8. Secondary Outcome: Recurrent or Progressive Malignancy
Description: Percentage of relapse estimated by cumulative incidence methods
Time Frame: At 12 months after the start of prednisone therapy
Measure: Number; unit: percentage of participants
Arm/Group | Group A (Low-dose) | Group B (Standard-dose)
Number analyzed (Participants) | 79 | 83
percentage of participants | 21 | 21

9. Secondary Outcome: Progression to Grade III-IV Acute GVHD
Description: Diagnosed and graded according to standard established criteria. Measure is percent of patients with baseline scores of IIa (Group A) or IIb (Group B) who progressed to more severe GVHD (Grade III/IV). Percentage estimated by cumulative incidence methods.
Time Frame: At approximately 100 days after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Group A (Low-dose) | Group B (Standard-dose)
Number analyzed (Participants) | 79 | 83
percentage of participants | 6 | 13
Statistical Analysis 1: Comparison: Group A (Low-dose) vs Group B (Standard-dose); Test type: Superiority or Other; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.14 to 1.33]

10. Secondary Outcome: Secondary Therapy for Acute GVHD Beyond Prednisone
Description: This includes any intervention intended to control acute GVHD through an immunosuppressive effect from oral or parenteral administration of any systemic medication not given previously. This does not include topical therapy, an increase in the dose of glucocorticoids or the resumption of treatment after previous discontinuation or any increase in the dose of immunosuppressive medication previously administered for GVHD prophylaxis, or reinstatement of GVHD prophylaxis previously discontinued. A change in treatment from cyclosporine to tacrolimus or vice versa because of drug toxicity is not considered secondary therapy, but any change made because of uncontrolled GVHD is considered secondary therapy. Percentage is estimated by cumulative incidence methods.
Time Frame: At approximately 100 days after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Group A (Low-dose) | Group B (Standard-dose)
Number analyzed (Participants) | 79 | 83
percentage of participants | 23 | 7
Statistical Analysis 1: Comparison: Group A (Low-dose) vs Group B (Standard-dose); Test type: Superiority or Other; p = 0.009, Regression, Cox; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.12 to 0.74]

11. Secondary Outcome: Chronic Extensive GVHD
Description: Percentage of patients with chronic extensive GVHD, estimated by cumulative incidence methods
Time Frame: At 12 months after the start of prednisone therapy
Measure: Number; unit: percentage of participants
Arm/Group | Group A (Low-dose) | Group B (Standard-dose)
Number analyzed (Participants) | 79 | 83
percentage of participants | 47 | 54

12. Secondary Outcome: Overall Survival
Description: Percentage of patients surviving as estimated by Kaplan-Meier.
Time Frame: At 12 months after the start of prednisone therapy
Measure: Number; unit: percentage of participants
Arm/Group | Group A (Low-dose) | Group B (Standard-dose)
Number analyzed (Participants) | 79 | 83
percentage of participants | 77 | 77
Statistical Analysis 1: Comparison: Group A (Low-dose) vs Group B (Standard-dose); Test type: Superiority or Other; p = 0.95, Regression, Cox; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.6 to 1.74]

ADVERSE EVENTS:
Description: Other (Non-serious) adverse events were not collected, only those events that could be caused by prednisone "under-treatment" were monitored. These include 1) the progression to grade III/IV acute GVHD, 2) the need for secondary systemic GVHD treatment, and 3) non-relapse mortality. These events are reported as secondary Outcome Measures.
Arm/Group | Arm I (Low-dose) | Arm II (Standard-dose)
Serious Adverse Events (participants affected / at risk) | 38/81 | 30/83
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Low-dose) (N=81) | Arm II (Standard-dose) (N=83)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
peripheral edema (Cardiac disorders) | 0 (0) | 1 (1)
palpitations (Cardiac disorders) | 1 (1) | 0 (0)
graft versus host disease (Immune system disorders) | 8 (9) | 0 (0)
lethargy (Nervous system disorders) | 0 (0) | 1 (1)
fever/infection (Infections and infestations) | 13 (14) | 11 (13)
orthostatic hypotension (Cardiac disorders) | 1 (1) | 0 (0)
gastroesophageal relux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
platelet infusion reaction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
relapse of hematological disease (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
suicide (Social circumstances) | 1 (1) | 0 (0)
adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
temporomandibular joint disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 1 (3) | 1 (1)
parotitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
mental status changes (Nervous system disorders) | 1 (1) | 2 (2)
hematopoietic graft failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
splenomagaly (Gastrointestinal disorders) | 0 (0) | 1 (1)
hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
elevated liver function tests (Hepatobiliary disorders) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 0 (0) | 1 (1)
leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
trauma/fall (General disorders) | 1 (1) | 0 (0)
weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
colonic pneumatosis (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes